CLINICAL TRIAL: NCT01047176
Title: Observational Prospective Study to esTIMAte the Rates of Outcomes in Patients Undergoing PCI With Drug Eluting Stent (DES) Implantation Who Take Statins
Brief Title: Observational Study to Estimate the Rates of Outcomes in Patients Undergoing Percutaneous Coronary Intervention (PCI) With Drug Eluting Stent (DES) Implantation Who Take Statins
Acronym: OPTIMA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CRU-CRE-2009/1
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Dyslipidemia; Coronary Heart Disease
Keywords: Statins; Coronary Heart Disease; Percutaneous coronary intervention (PCI)
MeSH Terms: conditions — Dyslipidemias; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Male or female > 18 year of age with indication to PCI

SUMMARY:
To estimate the rates of percutaneous coronary intervention (PCI) outcomes in patients after drug-eluting stents implantation who take statins.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina with indication to PCI
* Hospitalization to Russian Cardiological Research Center (РКНПК) for PCI procedure with drug-eluting stents implantation
* Statin therapy initiated for at least one month prior to PCI
* Written informed consent provided prior the start of participation in the study.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent.
* Presence of ACS during the current hospitalization
* Severe CHF (NYHA III/IV) or LVEF<40 %
* Stroke within 6 months before PCI
* Acute or chronic inflammatory disease
* Anti-inflammatory medications intake, with the exception of aspirin
* Severe liver or muscle disease
* Severe kidney disease / renal failure with creatinine > 3 mg/dl
* History of oncologic disease
* Conceivable impossibility to come in touch with the patient or his family at 1-year after the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patient
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To estimate the rates of percutaneous coronary intervention (PCI) outcomes in patients after drug-eluting stents implantation who take statins. | 3 visits for 12 month (before and after PCI)

SECONDARY OUTCOMES:
To evaluate prognostic factors (demographic, co-morbidity, smoking, LDL-C, inflammatory and cardiac markers) in patients undergoing PCI with drug eluting stent (DES) implantation who take statins and their association with PCI (MACCE) outcomes | 3 visits for 12 month
To estimate Low Density Lipoprotein Cholesterol (LDL-C) target level achievement and lipid-lowering therapy details in patients taking standard lipid lowering therapy prior the PCI. | 3 visits for 12 months
To estimate inflammatory markers (C-reactive protein (CRP) and Leukocytes) in patients prior and after PCI. | 3 visits for 12 months
To estimate cardiac markers (Troponin I, brain natriuretic peptide (BNP)) in patients before PCI. | 3 visits for 12 months
To study lipoprotein associated phospholipase A2 (Lp PLA2) in patients before PCI and its' association with PCI outcome. | 3 visits for 12 months
To study the rate of early and late stent thrombosis according to ARC classification | 3 visits for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuri A Karpov, Principal Investigator — RCRC (РКНПК)
Locations (1):
- Research Site, Moscow, Russia